CLINICAL TRIAL: NCT02442505
Title: Validation of the Modified Microlife Blood Pressure Monitor in Patients With Paroxysmal Atrial Fibrillation
Brief Title: Device-detected Paroxysmal Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: University of Birmingham (Other)
Collaborators: Sandwell & West Birmingham Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RG_13-114
Record Dates: First submitted 2015-05-01; First posted 2015-05-13 (Estimated); Last update posted 2019-04-19 (Actual); Status verified 2018-05

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Pacemaker; Device-detected; Sensitivity; Specificity
MeSH Terms: conditions — Atrial Fibrillation; Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Microlife WatchBP03 device — Microlife WatchBP03 device which is an automated oscillometric device using a new algorithm to detect atrial fibrillation

SUMMARY:
This study will use an automated blood pressure monitor (Microlife WatchBP03) with an inbuilt algorithm to detect atrial fibrillation (an irregular heart rhythm) in patients with an implanted pacemaker who have previously documented paroxysmal (intermittent) atrial fibrillation. This study will compare the Microlife device detected atrial fibrillation episodes to the pacemaker detected atrial fibrillation episodes.

DETAILED DESCRIPTION:
The modified Microlife blood pressure monitor is able to detect atrial fibrillation (AF) with high sensitivity (95%) and specificity (86%) and has a positive predictive value of 68% and negative predictive value of 98% for single readings. In addition, the modified device was also able to accurately classify the majority of the anomalous non-AF rhythms, although the specificity was highly variable, dependent upon the rhythm. However sinus rhythm was detected with a specificity of 97%. However, we do not currently know if the device would demonstrate a similar sensitivity in detecting AF in patients with paroxysmal AF.

Therefore, the present study will assess the sensitivity and specificity of the automated oscillometric device using a new AF algorithm among pacemaker patients with fast AF and atrial high-rate episodes and evaluate the effect of the specific rhythm abnormalities on the specificity for AF.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an implanted pacemaker for sick sinus syndrome with previously documented AF with atrial high-rate episodes

Exclusion Criteria:

* Any patient who's pacemaker has had previously documented atrial sensing or pacing problem issues
* Patients with permanent AF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have an implanted pacemaker for sick sinus syndrome with previously documented AF with atrial high-rate episodes, with be identified from the pacemaker clinic register at one NHS Trust. Patients with AF and one of the following pacemakers will be identified from this register: Medtronic Sensia DR, Medtronic Advisa DR, Sorin Reply DR, and St. Jude Medical Accent DR and the study population will be randomly drawn from these patients. Atrial high rate episodes will be defined as atrial rates ≥180 beats per minute [3-6]. The exclusion criteria will include any patient who's pacemaker has had previously documented atrial sensing or pacing problem issues and patients with permanent AF.
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2013-10; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who are identified as having atrial fibrillation by both the pacemaker and the Microlife device (%) | 24 hours
  True positive rate (sensitivity)
Percentage of patients who are identified as not having atrial fibrillation by both the pacemaker and the Microlife device (%) | 24 hours
  True negative rate (specificity)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory YH Lip, MD, Principal Investigator — University of Birmingham
Locations (1):
- Sandwell and West Birmingham Hospitals NHS Trust, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
IPD in an anonymised form can be made able upon direct request.